CLINICAL TRIAL: NCT06463574
Title: Evaluation of Micro -Tensile Bond Strength to Dentin and Color Stability of a New Self Adhesive Bulk-fill Resin Composite Restorative Material After Aging
Brief Title: Effect of Aging on Micro-tensile Bond Strength and Color Stability of Self-adhesive Resin Composite
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Minia University (Other)
Responsible Party: Principal Investigator, Nourhan Samir Soliman Ibrahim, Dr, Minia University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: self-adhesive resin composite
Record Dates: First submitted 2024-05-23; First posted 2024-06-18 (Actual); Last update posted 2024-06-18 (Actual); Status verified 2024-06

CONDITIONS: Tooth Decay
Keywords: Color stability; Aging; Self-adhesive
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Intervention Model Description: A total of 20 patients will be selected and divided randomly into two main groups according to the type of composite used, the first group will use Surefil one self-adhesive bulk-fill composite for restoring 10 posterior class I cavities and the second group will use 3M Filtek One high viscosity bulk-fill composite for restoring 10 posterior class I cavities.
Who Masked: Participant, Care Provider
Masking Description: This study is a prospective randomized clinical trial with a follow up of 6 months. The clinical examiner and the participant will be kept unaware of the treatment being administrated.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Surefil one bulk-fill composite (Experimental): Restorative material applied directly to the tooth without adhesive appliaction.
  Interventions: Other: self-adhesive resin restoration
- Filtek One bulk-fill composite (Active Comparator): Restorative material that is applied to the tooth after adhesive application.
  Interventions: Other: self-adhesive resin restoration

INTERVENTIONS:
Other: self-adhesive resin restoration — Light cured, hybrid resin composite material which contains polymerization modulator that lessens its degree of polymerization shrinkage
  Other Names: Surefil one

SUMMARY:
The objective of this study is to evaluate the micro-tensile bond strength of a newly self-adhesive resinous restorative material to dentin with and without application of universal bonding system (in-vitro) and to examine it's clinical performance by evaluation of it's color stability and marginal discoloration through a randomized clinical trial (in-vivo).

DETAILED DESCRIPTION:
For color stability and marginal discoloration test, twenty class I cavities were prepared in the molar teeth of twenty different patients and then were randomly divided into two groups of ten patients each, where half of the molars was restored with Surefil one self-adhesive bulk-fill composite and the other half with Filtek One bulk-fill composite. A VITA Easyshade spectrophotometer was used to measure the baseline color of the restoration and at the margin after 24 hours and degree of color change and marginal discoloration after 3 months and 6 months of composite placement and then degree of color change (ΔE) was determined using the CIE L*a*b* system. All discolored restored molar teeth of both composite types were polished using a series of different thickness of Sof-Lex aluminum oxide discs (coarse, medium, fine), then the degree of color change of the restoration and at the margin (ΔE) was determined and was then compared to the baseline color measurements.

ELIGIBILITY:
Inclusion Criteria:

* Patients with class I lesion in their maxillary or mandibular molars with a maximum of approximately 2 mm final cavity depth.
* Patients with teeth shade A2 according to Vitapan classical shade guide.
* Patients with an acceptable oral hygiene level.
* Patients keen to regularly attend the follow up visits.

Exclusion Criteria:

* Patients with heavy bruxism or traumatic occlusion.
* Patients with poor oral hygiene or active periodontal disease.
* Patients with exposed or endodontically treated teeth.
* Patients participated in a clinical trial within 6 months before beginning of this trial.
* Patients who decline to be involved in the study or sign the written consent.
* Patients unable to return for the follow up visits.

Ages: 25 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-06 (Estimated); Primary Completion 2024-11 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Clinical evaluation of color stability and marginal discoloration of resin restorations after aging in the patient mouth. | 6 months
  Clinical evaluation of degree of color change of resin restorations after aging in the patient mouth.

CONTACTS AND LOCATIONS:
Overall Officials: Wael Essam Jamil, Professor, Study Director — Faculty of Dental Medicine for Girls, AL-Azhar University
Locations (1):
- Faculty of Dentistry, Minya University., Minya, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Name Faculty Country
Supporting Information: Study Protocol
Time Frame: 6 months

REFERENCES:
- [Background] Ellithy MS, Abdelrahman MH, Afifi RR. Comparative clinical evaluation between self-adhesive and conventional bulk-fill composites in class II cavities: A 1-year randomized controlled clinical study. J Esthet Restor Dent. 2024 Sep;36(9):1311-1325. doi: 10.1111/jerd.13242. Epub 2024 Apr 24. PMID 38655672
- [Background] Rathke A, Pfefferkorn F, McGuire MK, Heard RH, Seemann R. One-year clinical results of restorations using a novel self-adhesive resin-based bulk-fill restorative. Sci Rep. 2022 Mar 10;12(1):3934. doi: 10.1038/s41598-022-07965-z. PMID 35273277
- [Background] Cieplik F, Scholz KJ, Anthony JC, Tabenski I, Ettenberger S, Hiller KA, Buchalla W, Federlin M. One-year results of a novel self-adhesive bulk-fill restorative and a conventional bulk-fill composite in class II cavities-a randomized clinical split-mouth study. Clin Oral Investig. 2022 Jan;26(1):449-461. doi: 10.1007/s00784-021-04019-y. Epub 2021 Jun 15. PMID 34129074
- [Background] Anwar RS, Hussein YF, Riad M. Optical behavior and marginal discoloration of a single shade resin composite with a chameleon effect: a randomized controlled clinical trial. BDJ Open. 2024 Feb 20;10(1):11. doi: 10.1038/s41405-024-00184-w. PMID 38378771
- [Background] Fidan M. The effects of different repolishing procedures on the color change of bulk-fill resin composites. Eur Oral Res. 2024 Jan 5;58(1):14-21. doi: 10.26650/eor.20231234627. PMID 38481725
- [Background] Uctasli MB, Garoushi S, Uctasli M, Vallittu PK, Lassila L. A comparative assessment of color stability among various commercial resin composites. BMC Oral Health. 2023 Oct 24;23(1):789. doi: 10.1186/s12903-023-03515-9. PMID 37875872